CLINICAL TRIAL: NCT05929131
Title: Video and Brochure and Discharge Instructions for Childhood Fever in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Aylin Kurt, assistant professor, Bartın Unıversity
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2022-SBB-0645
Record Dates: First submitted 2023-06-04; First posted 2023-07-03 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Fever; Child, Only
MeSH Terms: conditions — Fever | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- discharge instructions with video (Experimental): Parents who agree to participate in the study will be randomly assigned to the control or intervention groups. Before parents in the control group are discharged from the pediatric emergency service, a short 2-minute video will be shown to the American Academy of Pediatrics (2020) guidelines (intervention group with video) giving the same information about high fever to patients in addition to the verbal instructions. Instructions will be given by the same researcher to provide homogeneous and consistent information in all three groups. All patients will also receive a discharge report with instructions on post-treatment treatment.
  Interventions: Other: discharge instructions with video
- verbal discharge instructions only (Placebo Comparator): Parents who agree to participate in the study will be randomly assigned to the control or intervention groups. Parents in the control group will receive the usual verbal information and advice on high fever management in accordance with the guidelines of the American Academy of Pediatrics (2020) prior to discharge from the pediatric emergency service. Instructions will be given by the same researcher to provide homogeneous and consistent information in all three groups. All patients will also receive a discharge report with instructions on post-treatment treatment.
  Interventions: Other: verbal discharge instructions only
- discharge instructions with pamphlet (Experimental): Parents who agree to participate in the study will be randomly assigned to the control or intervention groups. Before the parents in the control group are discharged from the pediatric emergency service, in the second group (intervention group with brochure) in accordance with the guidelines of the American Academy of Pediatrics (2020), the parents will be told with the brochure giving the same information about fever in addition to the verbal instructions. Instructions will be given by the same researcher to provide homogeneous and consistent information in all three groups. All patients will also receive a discharge report with instructions on post-treatment treatment.
  Interventions: Other: discharge instructions with pamphlet

INTERVENTIONS:
Other: discharge instructions with pamphlet — Parents who agree to participate in the study will be randomly assigned to the control or intervention groups. Before the parents in the control group are discharged from the pediatric emergency service, in the second group (intervention group with brochure) in accordance with the guidelines of the American Academy of Pediatrics (2020), the parents will be told with the brochure giving the same information about fever in addition to the verbal instructions. Instructions will be given by the same researcher to provide homogeneous and consistent information in all three groups. All patients will also receive a discharge report with instructions on post-treatment treatment.
  Arms: discharge instructions with pamphlet
Other: discharge instructions with video — Parents who agree to participate in the study will be randomly assigned to the control or intervention groups. Before parents in the control group are discharged from the pediatric emergency service, a short 2-minute video will be shown to the American Academy of Pediatrics (2020) guidelines (intervention group with video) giving the same information about high fever to patients in addition to the verbal instructions. Instructions will be given by the same researcher to provide homogeneous and consistent information in all three groups. All patients will also receive a discharge report with instructions on post-treatment treatment.
  Arms: discharge instructions with video
Other: verbal discharge instructions only — Parents who agree to participate in the study will be randomly assigned to the control or intervention groups. Parents in the control group will receive the usual verbal information and advice on high fever management in accordance with the guidelines of the American Academy of Pediatrics (2020) prior to discharge from the pediatric emergency service. Instructions will be given by the same researcher to provide homogeneous and consistent information in all three groups. All patients will also receive a discharge report with instructions on post-treatment treatment.
  Arms: verbal discharge instructions only

SUMMARY:
This study was designed to evaluate whether adding Video discharge instructions to usual verbal information improves understanding of the information provided to caregivers of patients presenting to pediatric emergency departments for high fever. As secondary goals, it was aimed to assess whether video discharge instructions increase satisfaction with information received and reduce repeat visits.

DETAILED DESCRIPTION:
The research will be carried out in a randomized controlled manner. There will be three groups in the research: those who received video (intervention), brochure (intervention) and verbal (control) discharge instructions. A power analysis was performed based on the number of children in both groups, in another study in which the scales to be used in the research were used. According to the calculations made in the G-Power 3.1 Demo package program, when the effect size was accepted as 0.8, it was seen that at least 48 cases in each group would be sufficient for 80% power. Children who meet the research criteria will be assigned a random number to the intervention and control groups via http://www.randomize.org/ by numbering the order of arrival at the hospital. Research data will be collected using Descriptive Information Form and Parental Fever Management Scale and Post-Discharge Data Collection Form.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 1 month and 18 years old
* Parent's consent to participate in the research
* Parent's completion of all pre-and post-education follow-up

Exclusion Criteria:

* The child is not between 1 month and 18 years old
* The child does not undergo day surgery.
* Parent's refusal to participate in the research
* Parent not completing all pre- and post-education follow-up

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The parents in the groups who received discharge instructions with a video and brochure, three days later, had a lower "Parental Fever Management Scale" score average than the control group. | 3 days
  As a result of the answers given to the scale, the total score varies between 8 and 40. The increase in the total score of the scale indicates that parents developed high anxiety and fever phobia during the care of their children's febrile illnesses.

SECONDARY OUTCOMES:
The parents in the groups who received discharge instructions with a video and brochure, after three days, had higher scores on the "Fever Management Approach Scale" compared to the control group. | 3 days
  The scores that the participants can get vary between 6-36. Evaluation is defined as the participants with a score below 21 approaching the fire with fear, while the participants with a score above 20 contribute to fever management in children with a functional approach. Parents who receive discharge instructions with videos and brochures are expected to have an average score above 20.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartin Maternity and Pediatrics Hospital, Bartın, Turkey (Türkiye)

REFERENCES:
- [Derived] Kurt A, Dinc F, Gunes San E. Video and booklet discharge instructions for mothers for childhood fever in pediatric emergency department: A randomized controlled trial. Int Emerg Nurs. 2025 Feb;78:101546. doi: 10.1016/j.ienj.2024.101546. Epub 2024 Dec 4. PMID 39637747